CLINICAL TRIAL: NCT04355949
Title: Vitamin D, Vitamin B12, and Folic Acid Among Patients With Lifelong Premature Ejaculation and Non-responding to Dapoxetine Treatment.
Brief Title: Assessment of Serum Levels of Vitamin D, Vitamin B12 and Folic Acid Among Patients With Lifelong Premature Ejaculation and Non-responding to Dapoxetine Treatment.
Acronym: PE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohammed Abu El-Hamd, Assistant Professor of Dermatology, Venereology and Andrology Department, Faculty of Medicine, Sohag University, Egypt., Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2/2020
Record Dates: First submitted 2020-04-12; First posted 2020-04-21 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Vitamin D, Vitamin B12 and Folic Acid Among Patients With Premature Ejaculation
Keywords: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Intervention Model Description: assess serum levels of vitamin D, vitamin B12 and folic acid among patients with lifelong PE and non-responding to dapoxetine treatment.
Who Masked: Investigator
Masking Description: In a case-controlled clinical study, it will be carried out on 30 patients with lifelong PE and 30 healthy control subjects.
  Serum vitamin D, vitamin B12, and folic acid levels will be assessed in all subjects included in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with premature ejaculation (Experimental): Serum vitamin D, vitamin B12, and folic acid levels will be assessed
  Interventions: Diagnostic Test: Serum vitamin D, vitamin B12, folic acid
- Normal subjects (Experimental): Serum vitamin D, vitamin B12, and folic acid levels will be assessed
  Interventions: Diagnostic Test: Serum vitamin D, vitamin B12, folic acid

INTERVENTIONS:
Diagnostic Test: Serum vitamin D, vitamin B12, folic acid — Serum vitamin D, vitamin B12, and folic acid levels will be assessed
  Other Names: Serum vitamin D, vitamin B12, folic acid levels

SUMMARY:
Therefore, this study will aim to assess serum levels of vitamin D, vitamin B12 and folic acid among patients with lifelong PE and non-responding to dapoxetine treatment.

DETAILED DESCRIPTION:
We will consider the patients with LPE non-responding to dapoxetine treatment when they used the optimum dose (30 and 60mg) dapoxetine for 4 separate times with no response.

Serum vitamin D, vitamin B12, and folic acid levels will be assessed in all subjects included in the study. Venous blood samples will be drawn and kept into EDTA bottles in the morning between 8 and 10 a.m. after an overnight fast of about 10-14 hr.

ELIGIBILITY:
Inclusion Criteria:

* premature ejaculation
* non-responding to dapoxetine treatment.

Exclusion Criteria:

* diabetes mellitus,
* chronic prostatitis,
* Advanced renal or hepatic diseases
* neurological diseases and
* C.N.S. medications

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male patients with lifelong premature ejaculation and non-responding to dapoxetine treatment.
Enrollment: 60 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D in patient with PE | 0-1 week
  Serum vitamin D levels will be assessed Among Patients With Lifelong Premature Ejaculation and Non-responding to Dapoxetine Treatment.
vitamin B12, in patient with PE | 0-1 week
  vitamin B12 levels will be assessed Among Patients With Lifelong Premature Ejaculation and Non-responding to Dapoxetine Treatment.
folic acid in patient with PE | 0-1 week
  folic acid levels will be assessed Among Patients With Lifelong Premature Ejaculation and Non-responding to Dapoxetine Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Abu El-Hamd, MD, Principal Investigator — Dermatology, Venereology and Andrology, Faculty of Medicine, Sohag University
Locations (1):
- Faculty of Medicine, Sohag University, Egypt, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No